CLINICAL TRIAL: NCT03134092
Title: Life Stories for Opioid Risk Reduction in the ED
Brief Title: The Life STORRIED Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 826673
Record Dates: First submitted 2017-03-21; First posted 2017-04-28 (Actual); Results first posted 2020-08-17 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Opioid Dependence; Communication; Risk Behavior; Narrative Medicine
MeSH Terms: conditions — Opioid-Related Disorders; Communication; Risk-Taking; Narrative Medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Generalized Risk Communication (GRC) (No Intervention): Generalized Risk Communication (GRC): Participants in this arm will receive standard discharge instructions similar to instructions they would receive during usual care. This arm represents a standardized way of communicating post-discharge risk-benefit information about treatment options for patients with back pain and renal colic. The GRC, includes a standardized discharge information sheet about the clinical condition of interest and a written overview of population based evidence describing comparative benefits and side effects of alternative classes of medication acute pain.
- Probabilistic Risk Communication (PRT) (Active Comparator): Probabilistic Risk Communication (PRT): The probabilistic risk communication tool (PRT) is a visual tool that communicates risk using the previously validated Opioid Risk Tool (ORT). The ORT is designed to assess risk of opioid dependency for patients for whom an opioid pain relief prescription is being considered in outpatient settings. Patients in this arm will be given an iPad which will prompt them to take a short survey that automatically communicates their risk score. After which the iPad will show them a color coded visual thermometer that informs them of their risk of having issues related to opioids.
  Interventions: Other: Probabilistic Risk Communication Tool (PRT)
- Narrative Enhanced Risk Tool (NERT) (Active Comparator): Narrative Enhanced Risk Tool (NERT): Participants assigned to this arm will receive the PRT described above but will also be instructed to watch one or more narrative videos. This video intervention will include a brief narrative video of an individuals' cautionary tale related to prolonged opioid use. Narrative videos are developed from actual patient stories - put into a in a structured format of ~ 2-minute length and recorded.
  Interventions: Other: Probabilistic Risk Communication Tool (PRT); Other: Narrative Enhanced Risk Tool (NERT)

INTERVENTIONS:
Other: Probabilistic Risk Communication Tool (PRT) — The probabilistic risk communication tool (PRT) is a visual tool that communicates risk using the previously validated Opioid Risk Tool (ORT). The ORT is designed to assess risk of opioid dependency for patients for whom an opioid pain relief prescription is being considered in outpatient settings. Patients in this arm will be given an iPad which will prompt them to take a short survey that automatically communicates their risk score. After which the iPad will show them a color coded visual thermometer that informs them of their risk of having issues related to opioids.
  Arms: Narrative Enhanced Risk Tool (NERT); Probabilistic Risk Communication (PRT)
Other: Narrative Enhanced Risk Tool (NERT) — Participants assigned to this arm will receive the PRT described above but will also be instructed to watch one or more narrative videos. This video intervention will include a brief narrative video of an individuals' cautionary tale around prolonged opioid uses. Narrative videos are developed from actual patients sharing their stories - put into a in a structured format of ~ 2-minute length and recorded.
  Arms: Narrative Enhanced Risk Tool (NERT)

SUMMARY:
To compare the effectiveness of 3 strategies to inform patients of their risks associated with misuse of opioid prescriptions after treatment in the ED from renal colic or musculoskeletal back pain. Randomization will be to 3 arms for the Randomized Practical Control Trial across 3 sites (A) standardized general risk information sheet only (B) standardized general risk information sheet plus a visual probabilistic risk tool (C) standardized sheet plus narrative enhanced probabilistic risk tool.

DETAILED DESCRIPTION:
Amid a devastating public health crisis, in which 19,000 overdose deaths per year in the United States are due to prescription opioids, the investigators ask the following questions: Can risk-informed communication (with or without a narrative-enhanced tool) improve patient-centered outcomes in the domains of knowledge, opioid use, functional outcomes, and patient provider therapeutic alignment? This question has implications for over 17 million patients who present to acute care settings with acute pain from common conditions. Can these goals be accomplished in a real-world setting, for a diverse patient population? The investigators approach to this project includes a practical randomized controlled trial, conducted in nine acute care settings, at three geographically distinct hospital centers, with broad inclusion criteria and a diverse population. Aims: This project aims to compare the effectiveness of 1) a standardized general risk information sheet only; 2 a standardized general risk information sheet plus a probabilistic risk tool; and 3) a standardized sheet plus narrative-enhanced probabilistic risk tool on the following outcomes: * Knowledge as measured by risk awareness and treatment preferences for fewer opioids, particularly among those at higher risk for addiction * Reduced use of opioids as measured by quantity of opioids taken, functional improvement, and repeat use of unscheduled visits for pain at 14 days * Patient provider alignment as measured by concordance between patient preference and finalized prescription plan, and the presence of shared decision making. These aims will be achieved in a multicenter randomized practical clinical trial of 1,300 patients who are planned for discharge from acute care settings after being treated for acute back or acute kidney stone pain. The investigators hypothesize that, compared with patients receiving a generalized risk information sheet or a probabilistic risk communication tool alone, patients with acute renal colic and musculoskeletal back pain randomized to receive narrative-enhanced risk communication, will do the following: (H1) demonstrate greater knowledge, as determined by awareness of risk for opioid dependency; (H2a) select a treatment plan with fewer opioids; (H2b) take fewer opioids for fewer days, while achieving the same degree of pain relief and improved functional status; (H3a) enjoy greater levels of concordance between the patient-preferred and provider-selected treatment plans; and (H3b) engage in greater shared decision making with their providers. How these aims are important to patients: The research question is important to patients because 1) patients are frequently exposed to the potential for either under- or over-treatment of pain; 2) patients have different risk factors for dependency, which may impact the appropriateness of certain medications for pain relief; and 3) opioid dependence and misuse which often begin with prescriptions for acute pain are costly and common, and affect families, communities, and society as a whole.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years to 70 years old
* Experiencing back pain or renal colic
* Text messaging and internet access including email capabilities or access to a smartphone
* Anticipated discharge within 24 hours

Exclusion Criteria:

* Patients who take opioids for chronic pain or cancer treatments
* Patients who have taken opioids in the past month with the exception of patients who have taken opioids in the previous 48 hours before arriving at the ED for their presenting condition based on provider assessment
* Patients who are pregnant, in police custody, intoxicated, cognitively impaired, or otherwise unable to fully consent and participate
* Patients who are hemodynamically compromised, in respiratory distress, or in severe emotional or physical distress.
* Patients older than 70 or younger than 18
* Patients who will be admitted to hospital or deemed to have a critical illness based on provider assessment
* Patients who are cognitively impaired
* Patients who are suicidal or homicidal ideation by chart review and clinician assessment.
* Patients with evidence of aberrant behavior based on clinical assessment
* Patients who do not have a phone, text messaging OR email address
* Patients under police arrest at ED visit
* Patients who are non-English or Spanish speaking
* Patients previously enrolled
* Patient with any current contraindications for NSAIDs or opioid medications including allergies, chronic kidney disease (GFR60, if measured)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — If the patient identifies as male or female, we will enter that as such for the study.
Enrollment: 1302 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary F Meisel, MD, Principal Investigator — University of Pennsylvania
Locations (4):
- United States (4):
  - University of Alabama- Birmingham, Birmingham, Alabama
  - Mayo Clinic, Rochester, Minnesota
  - Northwell Health, Manhasset, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Meisel ZF, Shofer F, Dolan A, Goldberg EB, Rhodes KV, Hess EP, Bellamkonda VR, Perrone J, Cannuscio CC, Becker L, Rodgers MA, Zyla MM, Bell JJ, McCollum S, Engel-Rebitzer E, Tiako MJN, Ridgeway G, Schapira MM. A Multicentered Randomized Controlled Trial Comparing the Effectiveness of Pain Treatment Communication Tools in Emergency Department Patients With Back or Kidney Stone Pain. Am J Public Health. 2022 Feb;112(S1):S45-S55. doi: 10.2105/AJPH.2021.306511. PMID 35143273
- [Derived] Engel-Rebitzer E, Dolan AR, Aronowitz SV, Shofer FS, Nguemeni Tiako MJ, Schapira MM, Perrone J, Hess EP, Rhodes KV, Bellamkonda VR, Cannuscio CC, Goldberg E, Bell J, Rodgers MA, Zyla M, Becker LB, McCollum S, Meisel ZF. Patient Preference and Risk Assessment in Opioid Prescribing Disparities: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2021 Jul 1;4(7):e2118801. doi: 10.1001/jamanetworkopen.2021.18801. PMID 34323984
- [Derived] Meisel ZF, Goldberg EB, Dolan AR, Bansal E, Rhodes KV, Hess EP, Cannuscio CC, Schapira MM, Perrone J, Rodgers MA, Zyla MM, Bell JJ, McCollum S, Shofer FS. Stories to Communicate Individual Risk for Opioid Prescriptions for Back and Kidney Stone Pain: Protocol for the Life STORRIED Multicenter Randomized Clinical Trial. JMIR Res Protoc. 2020 Sep 24;9(9):e19496. doi: 10.2196/19496. PMID 32969832

RESULTS

PARTICIPANT FLOW:
Groups:
- Narrative Enhanced Risk Tool (NERT): Narrative Enhanced Risk Tool (NERT): Participants assigned to this arm will receive the PRT described above but will also be instructed to watch two narrative videos. This video intervention will include a brief narrative video of an individuals' experience with pain and/or pain treatment with opioids. Narrative videos were developed from actual patient stories - put into a in a structured format of ~ 2-minute length and recorded.
Period: Overall Study
Arm/Group | Generalized Risk Communication (GRC) | Probabilistic Risk Communication (PRT) | Narrative Enhanced Risk Tool (NERT)
Started | 434 | 435 | 433
Completed | 434 | 435 | 433
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Probabilistic Risk Communication (PRT): Probabilistic Risk Communication (PRT): The probabilistic risk communication tool (PRT) is a visual tool that communicates risk using the previously validated Opioid Risk Tool (ORT). The ORT is designed to assess risk of opioid dependency for patients for whom an opioid pain relief prescription is being considered in outpatient settings. Patients in this arm will be given an iPad which will prompt them to take a short survey that automatically communicates their risk score. After which the iPad will show them a color coded visual thermometer that informs them of their risk of having issues related to opioids.
  \
- Total: Total of all reporting groups
Arm/Group | Generalized Risk Communication (GRC) | Probabilistic Risk Communication (PRT) | Narrative Enhanced Risk Tool (NERT) | Total
Number analyzed (Participants) | 434 | 435 | 433 | 1302
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.2 (13.9) | 41.72 (16.6) | 40.32 (13.8) | 40.59 (13.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 224 | 229 | 239 | 692
  Male | 210 | 204 | 193 | 607
  Other | 0 | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/AA | 175 | 156 | 167 | 498
  White | 180 | 191 | 185 | 556
  Other/Multi-racial | 76 | 87 | 80 | 243
  Unknown | 3 | 1 | 1 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 434 | 435 | 433 | 1302
Educational Attainment [Count of Participants; unit: Participants]
  Less than high school | 29 | 25 | 31 | 85
  High School/GED | 131 | 117 | 137 | 385
  Some college/2-year degree | 137 | 139 | 119 | 395
  Bachelor's degree | 88 | 95 | 89 | 272
  Graduate or Professional school | 47 | 59 | 56 | 162
  Unknown | 2 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Risk Awareness and Recall
Description: The primary outcome of this study is for patients to gain an understanding of individual risk using the Opioid Risk Tool (ORT). The ORT is a brief screening tool allowing patients to confidentially enter their own history to determine the probability opioid dependency and addiction. High concordance between measured risk and patient recall might indicate sustained effectiveness (or stickiness) of the risk communication tool. Discordance might indicate a failure of risk communication and knowledge of individualized risk. This outcome is dichotomous, categorized as "Yes" the person correctly recalled their risk category or "No", either they did not correctly recall their risk category or they did not remember their risk category at all. The count of participants is the amount categorized as "Yes", they correctly recalled their risk category.
Time Frame: Day 14
Population: The control group was never made aware of their risk score as determined by the ORT. Additionally, there were participants who did not fill out the follow-up survey on Day 14, which is why their recall was not analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Probabilistic Risk Communication (PRT) | Narrative Enhanced Risk Tool (NERT)
Number analyzed (Participants) | 304 | 295
Participants | 118 | 129

2. Primary Outcome: Patient Reported Use of Opioid Medication
Description: Taking opioid medication at Day 14. This outcome is dichotomous. "Yes" if they were taking opioids at Day 14, or "No" if they were not taking opioids at Day 14.
Time Frame: Day 14
Population: There were some participants who did not complete the Day 14 survey, which is why not all participants were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Probabilistic Risk Communication (PRT): Probabilistic Risk Communication (PRT): The probabilistic risk communication tool (PRT) is a visual tool that communicates risk using the previously validated Opioid Risk Tool (ORT). The ORT is designed to assess risk of opioid dependency for patients for whom an opioid pain relief prescription is being considered in outpatient settings. Patients in this arm will be given an iPad which will prompt them to take a short survey that automatically communicates their risk score. After which the iPad will show them a color coded visual thermometer that informs them of their risk of having issues related to opioids.
  Probabilistic Risk Communication Tool (PRT): The probabilistic risk communication tool (PRT) is a visual tool that communicates risk using the previously validated Opioid Risk Tool (ORT). The ORT is designed to assess risk of opioid dependency for patients for whom an opioid pain relief prescription is being considered in outpatient settings. Patients in this arm will be given
- Narrative Enhanced Risk Tool (NERT): Narrative Enhanced Risk Tool (NERT): Participants assigned to this arm will receive the PRT described above but will also be instructed to watch one or more narrative videos. This video intervention will include a brief narrative video of an individuals' cautionary tale related to prolonged opioid use. Narrative videos are developed from actual patient stories - put into a in a structured format of ~ 2-minute length and recorded.
  Probabilistic Risk Communication Tool (PRT): The probabilistic risk communication tool (PRT) is a visual tool that communicates risk using the previously validated Opioid Risk Tool (ORT). The ORT is designed to assess risk of opioid dependency for patients for whom an opioid pain relief prescription is being considered in outpatient settings. Patients in this arm will be given an iPad which will prompt them to take a short survey that automatically communicates their risk score. After which the iPad will show them a color coded visual thermometer that infor
Arm/Group | Generalized Risk Communication (GRC) | Probabilistic Risk Communication (PRT) | Narrative Enhanced Risk Tool (NERT)
Number analyzed (Participants) | 317 | 301 | 294
Participants | 42 | 31 | 31

3. Secondary Outcome: Patient Reported Use of Opioid Medication
Description: A second outcome is measuring patient reported opioid medication use by Total morphine equivalents.
Time Frame: Days 1-2, days 4-6
Population: Data for this patient-reported outcome is not reliable. The question was not asked appropriately in order to accurately measure milligrams/dosage of prescription.
Arm/Group | Generalized Risk Communication (GRC) | Probabilistic Risk Communication (PRT) | Narrative Enhanced Risk Tool (NERT)
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Patient Reported Use of Opioid Medication
Description: Patient reported total pills taken in the first 48 hours after baseline enrollment.
Time Frame: Days 1-2
Measure: Count of Participants; unit: Participants
Groups:
- Narrative Enhanced Risk Tool (NERT): NERT: Participants assigned to this arm will receive the PRT described above but will also be instructed to watch one or more narrative videos. This video intervention will include a brief narrative video of an individuals' cautionary tale related to prolonged opioid use. Narrative videos are developed from actual patient stories - put into a in a structured format of ~ 2-minute length and recorded.
  Probabilistic Risk Communication Tool (PRT): The probabilistic risk communication tool (PRT) is a visual tool that communicates risk using the previously validated Opioid Risk Tool (ORT). The ORT is designed to assess risk of opioid dependency for patients for whom an opioid pain relief prescription is being considered in outpatient settings. Patients in this arm will be given an iPad which will prompt them to take a short survey that automatically communicates their risk score. After which the iPad will show them a color coded visual thermometer that informs them of their risk of having issues related to opioids.
  Narrative Enhanced Risk Tool (NERT): Participants assigned to this arm will receive the PRT described above but will also be instructed to watch one or more narrative videos. This video intervention will include a brief narrative video of an individuals' cautionary tale around prolonged opioid uses. Narrative videos are developed from actual patients sharing their stories - put into a in a structured format of ~ 2-minute length and recorded.
Arm/Group | Generalized Risk Communication (GRC) | Probabilistic Risk Communication (PRT) | Narrative Enhanced Risk Tool (NERT)
Number analyzed (Participants) | 243 | 243 | 242
Participants
  No opioids taken | 180 | 167 | 182
  1-2 opioid tablets taken | 35 | 26 | 26
  3-6 opioid tablets taken | 24 | 39 | 27
  >6 opioid tablets taken | 4 | 11 | 7

5. Secondary Outcome: Patient Reported Use of Opioid Medication
Description: Frequency of use
Time Frame: Day 14, 3 Months
Population: The number of participants analyzed differs from day 14 and day 90 because the total number analyzed is the number of participants still taking opioids at that time.
Measure: Count of Participants; unit: Participants
Arm/Group | Generalized Risk Communication (GRC) | Probabilistic Risk Communication (PRT) | Narrative Enhanced Risk Tool (NERT)
Number analyzed (Participants) | 42 | 31 | 31
Participants
  14 days: Daily | 13 | 19 | 13
  14 days: >3 times a week | 11 | 7 | 6
  14 days: 1-3 times a week | 10 | 2 | 6
  14 days: <1 time a week | 8 | 3 | 6
  90 days: number analyzed (Participants) | 24 | 19 | 16
  90 days: Daily | 9 | 5 | 4
  90 days: >3 times a week | 4 | 7 | 5
  90 days: 1-3 times a week | 5 | 2 | 4
  90 days: <1 time a week | 6 | 5 | 3

6. Secondary Outcome: Patient Reported Use of Opioid Medication
Description: Patient reported days to no longer taking opioids
Time Frame: Time from emergency department visit to ceasing opioid use. We assessed at days 1-2, 4-6, 14, and month 3, data up to 3 months reported.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Generalized Risk Communication (GRC) | Probabilistic Risk Communication (PRT) | Narrative Enhanced Risk Tool (NERT)
Number analyzed (Participants) | 164 | 162 | 148
Days | 6 [4 to 14] | 5 [4 to 14] | 4 [2 to 6]

7. Secondary Outcome: Reported Use of Non Opioid Pain Medication
Description: Patient reported use and dose of NSAIDs and acetaminophen
Time Frame: Days 1, day 14, 3 Months
Population: The number of participants analyzed changes at each time point based on the number of participants who filled out the surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | Generalized Risk Communication (GRC) | Probabilistic Risk Communication (PRT) | Narrative Enhanced Risk Tool (NERT)
Number analyzed (Participants) | 434 | 434 | 433
Participants
  Day 1: number analyzed (Participants) | 297 | 299 | 296
  Day 1: No pain medication | 47 | 55 | 64
  Day 1: NSAIDs only | 193 | 170 | 167
  Day 1: Opioids only | 15 | 20 | 16
  Day 1: Opioids and NSAIDs | 42 | 54 | 49
  Day 14: number analyzed (Participants) | 317 | 303 | 295
  Day 14: No pain medication | 144 | 142 | 147
  Day 14: NSAIDs only | 131 | 130 | 117
  Day 14: Opioids only | 15 | 11 | 8
  Day 14: Opioids and NSAIDs | 27 | 20 | 23
  Day 90: number analyzed (Participants) | 281 | 287 | 285
  Day 90: No pain medication | 154 | 163 | 171
  Day 90: NSAIDs only | 103 | 105 | 98
  Day 90: Opioids only | 9 | 9 | 3
  Day 90: Opioids and NSAIDs | 15 | 10 | 13

8. Secondary Outcome: Functional Ability/Return to Usual Activities
Description: The RAND health- 20 questionnaire will be used to measure functional ability. We report the domain of "Role Function".
  Scores for this domain are reported on a scale of 0% to 100%, with 0% representing the worst possible score in that domain and 100% the best possible score.
Time Frame: At Baseline and 3 Months (referred to as "3 M" below)
Population: Not all participants answered this question at both timepoints.
Measure: Least Squares Mean (95% Confidence Interval); unit: RAND Health score change baseline to 3 M
Arm/Group | Generalized Risk Communication (GRC) | Probabilistic Risk Communication (PRT) | Narrative Enhanced Risk Tool (NERT)
Number analyzed (Participants) | 434 | 434 | 433
RAND Health score change baseline to 3 M | 5.45 [1.29 to 9.62] | 5.10 [1.01 to 9.20] | 4.26 [0.14 to 8.37]

9. Secondary Outcome: Functional Ability/Return to Usual Activities
Description: The American Pain Outcome questionnaire will be used to measure functional ability. We report the change in the score for "In the last 24 hours how much has pain interfered/prevented you from... Doing activities such as walking, sitting, or standing" between Baseline and 3 months. (scale: 0 = 0% of the time, 10 = 100% of the time)
Time Frame: Baseline, Days 1 and 7, Day 14, 3 Months (referred to as "3 M" below)
Population: Not all participants answered the question at both time points.
Measure: Least Squares Mean (95% Confidence Interval); unit: APO score change baseline to 3 M
Groups:
- Narrative Enhanced Risk Tool (NERT): Narrative Enhanced Risk Tool (NERT): Participants assigned to this arm will receive the PRT but will also be instructed to watch one or more narrative videos. This video intervention will include a brief narrative video of an individuals' cautionary tale related to prolonged opioid use. Narrative videos are developed from actual patient stories - put into a in a structured format of ~ 2-minute length and recorded.
  Probabilistic Risk Communication Tool (PRT): The probabilistic risk communication tool (PRT) is a visual tool that communicates risk using the previously validated Opioid Risk Tool (ORT). The ORT is designed to assess risk of opioid dependency for patients for whom an opioid pain relief prescription is being considered in outpatient settings. Patients in this arm will be given an iPad which will prompt them to take a short survey that automatically communicates their risk score. After which the iPad will show them a color coded visual thermometer that informs them of their risk of having issues related to opioids.
  Narrative Enhanced Risk Tool (NERT): Participants assigned to this arm will receive the PRT described above but will also be instructed to watch one or more narrative videos. This video intervention will include a brief narrative video of an individuals' cautionary tale around prolonged opioid uses. Narrative videos are developed from actual patients sharing their stories - put into a in a structured format of ~ 2-minute length and recorded.
Arm/Group | Generalized Risk Communication (GRC) | Probabilistic Risk Communication (PRT) | Narrative Enhanced Risk Tool (NERT)
Number analyzed (Participants) | 434 | 434 | 433
APO score change baseline to 3 M | 4.46 [3.69 to 5.23] | 4.82 [4.06 to 5.59] | 4.67 [3.70 to 5.24]

10. Secondary Outcome: Patient Reported Shared Decision Making
Description: The CollaboRATE93 scale- a brief, patient reported measure of shared decision making after a clinical encounter will be used. The scale will be adapted to reflect the context of an acute pain clinical encounter in the emergency department. There are three questions scored 0-9 with higher values meaning more collaboration. The average score of the three questions was calculated.
Time Frame: Day 1
Population: There were participants that did not fill out the Day 1 survey and were therefore not analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Generalized Risk Communication (GRC) | Probabilistic Risk Communication (PRT) | Narrative Enhanced Risk Tool (NERT)
Number analyzed (Participants) | 306 | 310 | 310
score on a scale | 6.826797 [6.566200 to 7.0873951] | 7.070968 [6.812057 to 7.3298782] | 7.220430 [6.961520 to 7.4793413]

11. Secondary Outcome: Satisfaction With Pain Treatment
Description: Participants are asked "How satisfied were you with the results of your pain treatment while in the hospital?" with 0 = extremely dissatisfied and 10 = extremely satisfied.
Time Frame: Days 1 and 7, Day 14, 3 Months
Population: A different number of participants filled out the surveys at each time point. Therefore, the number above, overall participants analyzed, reflects the overall numbers randomized to each arm.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Generalized Risk Communication (GRC) | Probabilistic Risk Communication (PRT) | Narrative Enhanced Risk Tool (NERT)
Number analyzed (Participants) | 434 | 435 | 433
score on a scale
  Day 1: number analyzed (Participants) | 307 | 309 | 308
  Day 1 | 6.57 [6.21 to 6.93] | 6.58 [6.22 to 6.94] | 7.25 [6.89 to 7.61]
  Day 7: number analyzed (Participants) | 300 | 298 | 296
  Day 7 | 6.50 [6.12 to 6.88] | 6.49 [6.11 to 6.87] | 6.92 [6.54 to 7.30]
  Day 14: number analyzed (Participants) | 315 | 302 | 296
  Day 14 | 6.58 [6.20 to 6.96] | 6.56 [6.17 to 6.95] | 6.82 [6.43 to 7.21]
  Month 3: number analyzed (Participants) | 282 | 285 | 282
  Month 3 | 6.58 [6.18 to 6.98] | 6.81 [6.41 to 7.21] | 7.17 [6.77 to 7.57]

12. Secondary Outcome: Trust in Provider
Description: The Trust in Physician scale, will be used to measure the patient's their trust in their provider. Allows Patient to report their perception of their provider. Patients are more likely to be adherent to medical care when they trust their physicians. We report the "Trust in lead clinician" item. Score 0-100, where higher indicates more trust.
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Generalized Risk Communication (GRC) | Probabilistic Risk Communication (PRT) | Narrative Enhanced Risk Tool (NERT)
Number analyzed (Participants) | 300 | 298 | 296
score on a scale | 76.23 (21.91) | 73.62 (23.93) | 75.20 (21.06)

13. Secondary Outcome: Patient Preference for Treatment Plan
Description: Patients will be provided options for pain treatment for discharge treatment plan. We are reporting out on patients who indicated they preferred any type of opioid.
Time Frame: At Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Generalized Risk Communication (GRC) | Probabilistic Risk Communication (PRT) | Narrative Enhanced Risk Tool (NERT)
Number analyzed (Participants) | 434 | 434 | 432
Participants | 143 | 123 | 112

14. Secondary Outcome: Treatment Plan Agreement Between Patient Preference and Provider Decision
Description: Patient preference will be linked to electronic medical record data. Discordance between risk informed patient preferences and provider selection may indicate failure to achieve an optimized patient centered outcome. We report overall alignment.
Time Frame: At Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Generalized Risk Communication (GRC) | Probabilistic Risk Communication (PRT) | Narrative Enhanced Risk Tool (NERT)
Number analyzed (Participants) | 434 | 433 | 432
Participants | 286 | 300 | 303

15. Secondary Outcome: Self-Report Additional Provider Visits
Description: Self-Report additional provider visits to measure follow-up visits for pain
Time Frame: Day 14 and 3 Month
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Generalized Risk Communication (GRC) | Probabilistic Risk Communication (PRT) | Narrative Enhanced Risk Tool (NERT)
Number analyzed (Participants) | 434 | 434 | 433
Participants
  Day 14: number analyzed (Participants) | 317 | 302 | 295
  Day 14 | 125 | 127 | 121
  Day 90: number analyzed (Participants) | 281 | 287 | 286
  Day 90 | 113 | 128 | 124

16. Secondary Outcome: Current Opioid Misuse Measure (COMM)
Description: The Current Opioid Misuse measure (COMM) will be used to measure misuse of opioids.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Generalized Risk Communication (GRC) | Probabilistic Risk Communication (PRT) | Narrative Enhanced Risk Tool (NERT)
Number analyzed (Participants) | 24 | 19 | 16
Participants | 17 | 9 | 9

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 4 months.
Description: The study team did not track mortality or specific adverse events, as there were no reasonable expectations that our communication interventions would impact mortality.
Arm/Group | Generalized Risk Communication (GRC) | Probabilistic Risk Communication (PRT) | Narrative Enhanced Risk Tool (NERT)
All-Cause Mortality (participants affected / at risk) | 0/434 | 0/435 | 0/433
Serious Adverse Events (participants affected / at risk) | 0/434 | 0/435 | 0/433
Other Adverse Events (participants affected / at risk) | 0/434 | 0/435 | 0/433

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT03134092/Prot_SAP_001.pdf